CLINICAL TRIAL: NCT03417479
Title: Gabapentin Premedication for Pediatric Anterior Cruciate Ligament Reconstruction: Randomized Control Trial
Brief Title: Gabapentin Premedication for ACL Reconstruction: RCT
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: CHOA IRB 15-094
Record Dates: First submitted 2017-09-26; First posted 2018-01-31 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2019-07

CONDITIONS: Anterior Cruciate Ligament (ACL) Reconstruction
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1:1 Randomization: Patients will be randomized to either a single dose of 15mg/kg up to 600 mg of gabapentin or a placebo equivalent at a 1:1 ratio. The subjects will be enrolled in the study at the orthopedic surgeon's office with randomization occurring on the day of surgery by the hospital pharmacist. The method for the randomization will be the creation of a sequence of sealed envelopes containing assignment information for a dose of 600 mg of gabapentin or placebo.
  Interventions: Other: Gabapentin

INTERVENTIONS:
Other: Gabapentin
  Other Names: Neurontin

SUMMARY:
This double blind randomized control trial will enroll 100 participants ages 12-18 years, undergoing ACL repair. Participants receive gabapentin or placebo preoperatively. Outcome measurements of self-reported pain score using scale of 1 to 10 with 10 being the worse obtained from the EMR and participants interviews with a phone nurse for five days postoperatively to determine severity of pain as well as use of opioids.

DETAILED DESCRIPTION:
Anterior Cruciate Ligament (ACL) injury and surgical repair occurs in 200,000 active adolescent and young adult patients each year. ACL repair is associated with significant postoperative pain. Current methodologies for pain include regional nerve blocks, opioid or non-steroidal analgesia. Few studies have evaluated use of neuro-inhibitors such as gabapentin to limit pain response.

The purpose of this study then is to examine the use of gabapentin in reducing postoperative pain in adolescent ACL patients. The investigators hypothesize one 15mg/kg (up to 600mg) dose of gabapentin preoperatively would reduce: 1) self-reported postoperative pain and, 2) opioid use compared to patients who do not receive preoperative gabapentin.

This double blind randomized control trial will enroll 100 participants ages 12-18 years, undergoing ACL repair. Participants receive gabapentin or placebo preoperatively. Outcome measurements of self-reported pain score using scale of 1 to 10 with 10 being the worse obtained from the EMR and participant interviews with a phone nurse for five days postoperatively to determine severity of pain as well as use of opioids.

Outcome measurements will give a more comprehensive description of the postoperative experience and test gabapentin's opioid sparing effect. Due to paucity of literature on pain relief in this population, this pilot study will inform a larger multi-site study.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification 1 or 2
* Scheduled for elective ACL surgery in pediatric outpatient setting

Exclusion Criteria:

* BMI greater than 40
* ASA classification greater than 2
* Recurrent ACL reconstruction
* Allograft ACL reconstruction
* History of renal insufficiency
* History of chronic pain
* Allergy to Gabapentin

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Inclusion criteria include patients ages 12-18 years with an ASA class 1 or 2 scheduled for elective ACL reconstruction in the outpatient setting by Dr. Michael Busch. Exclusion criteria include a BMI >40, recurrent ACL reconstruction, allograft ACL reconstruction, history of renal insufficiency, chronic pain or allergy to gabapentin.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Effective Dose determination | 5 days post surgery
  To determine whether one 15mg/kg (up to 600 mg) dose of gabapentin preoperatively reduces pain after ACL surgery over the first 5 days of the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Gettis, DNP, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gettis M, Brown AM, Fujimoto A, Wetzel M, Thomsen J. Gabapentin Premedication to Reduce Postoperative Pain for Pediatric Tonsillectomy/Adenoidectomy: A Pilot Study. J Perianesth Nurs. 2022 Oct;37(5):626-631. doi: 10.1016/j.jopan.2021.11.011. Epub 2022 Mar 5. PMID 35256248